CLINICAL TRIAL: NCT01550432
Title: Effects of GSH and N-Acetylcysteine on Inflammatory Markers Among Adults With CVD Risk
Brief Title: Effects of Glutathione (an Antioxidant) and N-Acetylcysteine on Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Christopher Gardner, Associate Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SU-03252010-5442; R21AT004475 (NIH)
Record Dates: First submitted 2011-06-27; First posted 2012-03-12 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Obesity; Hyperlipidemia; Insulin Resistance; Hypertension
MeSH Terms: conditions — Obesity; Hyperlipidemias; Insulin Resistance; Hypertension | interventions — Glutathione; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- High-Dose Glutathione (Experimental): 2,260 mg/day
  Interventions: Dietary Supplement: Glutathione
- Low-Dose Glutathione (Experimental): 1,130 mg/day
  Interventions: Dietary Supplement: Glutathione
- High-Dose N-Acetylcysteine (Experimental): 1,200 mg/day
  Interventions: Dietary Supplement: N-Acetylcysteine
- Low-Dose N-Acetylcysteine (Experimental): 600 mg/day
  Interventions: Dietary Supplement: N-Acetylcysteine
- Placebo (Placebo Comparator): Volume of liquid placebo product comparable to glutathione and 1 or 2 placebo pills/day.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Glutathione — 1,130 mg/day or 2,260 mg/day for 8 weeks
  Other Names: ReadiSorb
  Arms: High-Dose Glutathione; Low-Dose Glutathione
Dietary Supplement: N-Acetylcysteine — 600 mg/day or 1,200 mg/day for 8 weeks
  Other Names: Twinlab
  Arms: High-Dose N-Acetylcysteine; Low-Dose N-Acetylcysteine
Other: Placebo — Volume of liquid placebo product comparable to liposomal glutathione and 1 or 2 placebo pills/day.
  Other Names: Nutrilite
  Arms: Placebo

SUMMARY:
The rationale for the potential role of antioxidants in the prevention of cardiovascular diseases (CVD) remains strong despite the disappointing results of recent trials with a few select antioxidant vitamins. Glutathione (GSH) is one of the body's most powerful antioxidant agents but there is a surprising paucity of data on its use as an interventional therapy.

Glutathione, when taken orally, is immediately broken down into its constituent amino acids, of which cysteine is the only one to be essential. Available cysteine is the critical determinant of intracellular GSH concentrations. N-acetyl cysteine (NAC) is an antioxidant supplement that has been used to provide a source of cysteine to replete GSH levels. By replenishing endogenous glutathione, it is possible that NAC would exert the same effect(s) as exogenous GSH.

However, there is a new delivery system, liposomal GSH, which keeps glutathione intact. In this study, the investigators propose to match the cysteine content of NAC and GSH and compare the effects of these two supplements, at two different doses, on markers of inflammation and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: Both women and men
2. Age: > or = 18 years
3. Ethnicity and race: All ethnic and racial backgrounds welcome
4. Presence of Metabolic Syndrome: As defined in ATP III of the National 5.Cholesterol Education program, the metabolic syndrome will be diagnosed as presence of at least three of the following, which will be measured at the screening clinic visit:

   * Central obesity as measured by waist circumference:

     * Men: Greater than 40 inches
     * Women: Greater than 35 inches
   * Fasting blood triglycerides greater than or equal to 150 mg/dL
   * Blood HDL cholesterol:

     * Men: Less than 40 mg/dL
     * Women: Less than 50 mg/dL
   * Blood pressure greater than or equal to 130/85 mmHg
   * Fasting glucose greater than or equal to 100 mg/dL

6.Planning to be available for clinic visits and bottle pick-ups for the 8 weeks of study participation 7.Ability and willingness to give written informed consent 8.No known active psychiatric illness.

Exclusion Criteria:

1. Daily intake of dietary supplements containing antioxidants or omega-3 FAs
2. Fasting blood glucose > 140 mg/dL
3. Significant liver enzyme abnormality

   * AST or ALT more than 2 times the upper limit of normal and/or
   * Bilirubin more than 50% the upper limit of normal
   * Renal disease as measured at baseline:
   * Serum creatinine > 1.30 mg/dL, or
   * Calculated creatinine clearance < 71 mL/min
4. Self reported personal history of:

   * Clotting disorders
   * Clinically significant atherosclerosis (e.g., CAD, PAD)
   * Malignant neoplasm
   * Ongoing infection
   * Inflammatory disease (e.g., rheumatoid arthritis)
5. Subjects currently receiving the following medications (self report):

   * Anti-Inflammatory drugs
   * Lipid lowering drugs including statins
   * Anti-hypertensive drugs
   * Anti-coagulant drugs
6. Body Mass Index (BMI) greater than or equal to 40.
7. Pregnant or Lactating
8. Inability to communicate effectively with study personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Inflammatory Markers | 8 weeks

SECONDARY OUTCOMES:
Oxidized LDL | 8 weeks
Insulin Sensitivity | 8 weeks
Weight | 8 weeks
Blood pressure | 8 weeks
Serum lipids | 8 weeks
Insulin | 8 weeks
Glucose | 8 weeks
Plasma Glutathione levels | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Gardner, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No